CLINICAL TRIAL: NCT01042639
Title: The Effect of Physical Activity on Bone Strength and Immune System in Very Low Birth Weight Infants: is More Really Better??
Brief Title: The Effect of Physical Activity on Bone Mineralization and Immune System in Very Low Birth Weight Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 060-09
Record Dates: First submitted 2009-12-31; First posted 2010-01-05 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Osteopenia of Prematurity
Keywords: osteopenia; very low birthweight infants; bone speed of sound; quantitative ultrasound
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- physical activity once a day (Active Comparator)
  Interventions: Behavioral: passive physical activity
- physical activity twice a day (Experimental)
  Interventions: Behavioral: passive physical activity
- control (No Intervention)
  Interventions: Behavioral: passive physical activity

INTERVENTIONS:
Behavioral: passive physical activity — extension and flexion range-of-motion exercise against passive resistance of both the upper and lower extremities. Both extension and flexion were performed five times at the wrist, elbow, shoulder, ankle, knee, and hip joints
  Other Names: passive range-of-motion exercise against passive resistance.

SUMMARY:
Studies have demonstrated that brief (5-10 min a day) passive range-of-motion exercise is beneficial for bone development in very low birth weight (VLBW) preterm infants. However, the optimal duration and frequency of exercise for bone development in preterm infants is yet unknown.

The effect of exercise on the immune system was widely studied in adult and children. Exercise induces increase in IL-6, IL-10, and IL1ra. In adult even 10 minutes of flexion and extension of the wrist cause systemic increase in IL-6. The effect of physical activity on pro and anti inflammatory cytokines in preterm infant was not studied.

Objectives:

1. To assess weather twice daily exercise intervention will enhance bone strength compared to once a day intervention
2. To evaluate the effect of a single exercise intervention on inflammatory mediators.

Methods:

Single center (Meir Medical Center), double blind, randomized control study.

DETAILED DESCRIPTION:
Infants will be randomly assigned to one of 3 study groups. Group 1 - physical activity once a day. Group 2 - physical activity twice a day and group 3 - control.

The physical activity program is based on the Moyer-Mileur et al protocol (1). Briefly, this protocol involves extension and flexion range-of-motion exercise against passive resistance of both the upper and lower extremities. Both extension and flexion were performed five times at the wrist, elbow, shoulder, ankle, knee, and hip joints (about 10 minutes for each session). Infant in group 1 have the physical activity intervention once a day, 5 days a week. Infant in group 2 will have the same physical activity intervention twice a day, five times a week. Infant in group 3, the control group will have a similar time (10 minutes) of daily interactive periods of holding and stroking without range-of-motion activity.

The physical activity will be done by the same person (the NICU physiotherapist) Growth parameters, and bone strength, will be measured at enrollment and every 2 weeks till discharge.

Bone strength assessment will be determined by quantitative ultrasound measurement of bone speed of sound (SOS) at the middle left tibial shaft (Sunlight Omnisense Premier). All measurements will be performed by the same person, who will be blinded to the group assignment.

Cytokines study In a sub-group of patients who will have arterial line at enrollment blood sample ( 0.6 CC) will be drawn before and immediately following activity for assessment of proinflammatory (IL-6) and anti-inflammatory ( IL1-ra) cytokines. Samples will be kept at -20º C and will be analyzed after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight<1500gr, appropriate for gestational age.
2. After initial cardio-respiratory stabilization
3. < 14 days postnatal age
4. Written parental informed consent

Exclusion Criteria:

1. Intrauterine growth retardation
2. Severe central nervous system disorder (including IVH grade 3-4).
3. Congenital anomalies/chromosomal abnormalities.
4. Congenital bone disease.

Ages: 3 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Bone Speed of sound | during hospitalization

SECONDARY OUTCOMES:
Anthropometric measurements | During hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ita Litmanovitz, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Moyer-Mileur L, Luetkemeier M, Boomer L, Chan GM. Effect of physical activity on bone mineralization in premature infants. J Pediatr. 1995 Oct;127(4):620-5. doi: 10.1016/s0022-3476(95)70127-3. PMID 7562289